CLINICAL TRIAL: NCT02208245
Title: Prospective Randomized Clinical Trial Comparing Infraclavicular Versus Axillary Approach to Brachial Plexus Block.
Brief Title: Prospective Clinical Trial Comparing Infraclavicular Versus Axillary Approach to Brachial Plexus Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Leonardo Henrique Cunha Ferraro, MD, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Infra Study
Record Dates: First submitted 2014-07-30; First posted 2014-08-05 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-08

CONDITIONS: Scaphoid Fractures; Distal Radius Fractures; Wrist Injury Arthrodesis
MeSH Terms: conditions — Wrist Fractures | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultrasound: Axillary block (Active Comparator): For the axillary group, the ultrasound probe will be placed upright in the armpit to obtain a cross section of this region. After visualization of the nerves form the brachial plexus by ultrasound, 5 mL of ropivacaine 0.5% will be injected around each nerve to be blocked (median, ulnar, radial and musculocutaneous). If resistance to the injection of the solution is present or the patient complains of severe pain, the needle will be immediately repositioned.
  Interventions: Device: Ultrasound: Axillary block; Drug: Ropivacaine
- Ultrasound: Infraclavicular block (Active Comparator): For the infraclavicular group, the ultrasound probe will be placed in the infraclavicular region (the junction between the clavicle and the coracoid process) to obtain a cross-sectional imaging of the axillary artery. After visualization of the axillary artery by ultrasound, the block will be performed using the technique in plan for visualization of the needle. The needle is placed in position 6-8 hours of the artery, and 20 mL of ropivacaine 0.5% will be injected, observing a dispersal of local anesthetic around the artery.
  Interventions: Device: Ultrasound: Infraclavicular block; Drug: Ropivacaine

INTERVENTIONS:
Device: Ultrasound: Axillary block — Ultrasound guided axillary block
  Arms: Ultrasound: Axillary block
Device: Ultrasound: Infraclavicular block — Ultrasound guided infraclvicular block
  Arms: Ultrasound: Infraclavicular block
Drug: Ropivacaine — 20 ml of ropivacaine 0,5% in both groups ( axillary block and infraclavicular block)

SUMMARY:
The brachial plexus block is an anesthetic technique often used for surgical procedures of the upper limb. To get the brachial plexus block, several routes can be used, including the axillary and infraclavicular approach.

Few studies have compared these techniques, considering the time to perform the block, the onset time and success rate, with conflicting results. Furthermore, there is little information in the literature comparing the length of postoperative analgesia provided by these techniques.

Therefore, the investigators designed this study in order to elucidate the differences between these two techniques to assist the anesthesiologist to choose the best of them in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* age older than 18 years and less than 70 years
* consent informed signed by the patient
* candidates for surgical intervention of scaphoid fractures, distal radius fractures and wrist arthrodesis
* American Society of Anesthesiology physical status I, II and III
* body mass index (BMI) <35 kg / m².

Exclusion Criteria:

* cognitive impairment or active psychiatric condition
* infection at the puncture site
* bleeding disorders
* history of allergy to ropivacaine

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2014-02; Primary Completion 2015-03 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
postoperative analgesia | first postoperative day
  All patients will be contacted on the first postoperative day to tell the time of onset of pain postoperatively. The duration of postoperative analgesia is defined as the interval between the end of local anesthetic injection and the onset of postoperative pain reported by the patient.

SECONDARY OUTCOMES:
local anesthetic pharmacokinetics | During the procedure
  Venous blood samples will be taken from some patients through a cannula. The samples will be used for the determination of serum levels achieved after ropivacaine blockade. Samples will be taken every 15 minutes during the first hour, every 30 minutes during the second hour and 4 hours after the blockade. These samples will be analyzed using the technique of high performance liquid chromatography coupled with mass spectrometry.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Angela Tardelli, PhD, Study Director — Federal University of São Paulo
Locations (1):
- Federal University of Sao Paulo - Hospital Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Tran DQ, Russo G, Munoz L, Zaouter C, Finlayson RJ. A prospective, randomized comparison between ultrasound-guided supraclavicular, infraclavicular, and axillary brachial plexus blocks. Reg Anesth Pain Med. 2009 Jul-Aug;34(4):366-71. doi: 10.1097/AAP.0b013e3181ac7d18. PMID 19574871
- [Background] Song IA, Gil NS, Choi EY, Sim SE, Min SW, Ro YJ, Kim CS. Axillary approach versus the infraclavicular approach in ultrasound-guided brachial plexus block: comparison of anesthetic time. Korean J Anesthesiol. 2011 Jul;61(1):12-8. doi: 10.4097/kjae.2011.61.1.12. Epub 2011 Jul 21. PMID 21860745
- [Background] Lopez-Morales S, Moreno-Martin A, Leal del Ojo JD, Rodriguez-Huertas F. [Ultrasound-guided axillary block versus ultrasound-guided infraclavicular block for upper extremity surgery]. Rev Esp Anestesiol Reanim. 2013 Jun-Jul;60(6):313-9. doi: 10.1016/j.redar.2013.02.012. Epub 2013 May 15. Spanish. PMID 23684374
- [Background] Koscielniak-Nielsen ZJ, Frederiksen BS, Rasmussen H, Hesselbjerg L. A comparison of ultrasound-guided supraclavicular and infraclavicular blocks for upper extremity surgery. Acta Anaesthesiol Scand. 2009 May;53(5):620-6. doi: 10.1111/j.1399-6576.2009.01909.x. PMID 19419356
- [Background] Ootaki C, Hayashi H, Amano M. Ultrasound-guided infraclavicular brachial plexus block: an alternative technique to anatomical landmark-guided approaches. Reg Anesth Pain Med. 2000 Nov-Dec;25(6):600-4. doi: 10.1053/rapm.2000.18184. PMID 11097667
- [Background] Sandhu NS, Capan LM. Ultrasound-guided infraclavicular brachial plexus block. Br J Anaesth. 2002 Aug;89(2):254-9. doi: 10.1093/bja/aef186. PMID 12378663
- [Background] Tran DQ, Clemente A, Tran DQ, Finlayson RJ. A comparison between ultrasound-guided infraclavicular block using the "double bubble" sign and neurostimulation-guided axillary block. Anesth Analg. 2008 Sep;107(3):1075-8. doi: 10.1213/ane.0b013e31817ef259. PMID 18713932
- [Background] Arcand G, Williams SR, Chouinard P, Boudreault D, Harris P, Ruel M, Girard F. Ultrasound-guided infraclavicular versus supraclavicular block. Anesth Analg. 2005 Sep;101(3):886-890. doi: 10.1213/01.ANE.0000159168.69934.CC. PMID 16116009
- [Background] Ferraro LH, Takeda A, dos Reis Falcao LF, Rezende AH, Sadatsune EJ, Tardelli MA. Determination of the minimum effective volume of 0.5% bupivacaine for ultrasound-guided axillary brachial plexus block. Braz J Anesthesiol. 2014 Jan-Feb;64(1):49-53. doi: 10.1016/j.bjane.2013.03.014. Epub 2013 Dec 2. PMID 24565388